CLINICAL TRIAL: NCT04255459
Title: Post-Market Surveillance of Tobacco Products: A Multicenter Clinical Trial of Natural Adopters of Cigarettes, Moist Snuff, Camel SNUS, and Dual Use
Brief Title: Post-Market Surveillance of Tobacco Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSD0904
Record Dates: First submitted 2019-09-04; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Smoking, Tobacco; Smoking Behaviors
MeSH Terms: conditions — Tobacco Smoking; Smoking | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Moist Snuff users (Other): Subjects for whom moist snuff is their usual brand of tobacco product.
  Interventions: Other: Moist Snuff
- Camel Snus users (Other): Subjects for whom Camel Snus is their usual brand of tobacco product.
  Interventions: Other: Camel Snus
- Dual users of Camel Snus and cigarette (Other): Subjects who use both Camel Snus and cigarettes as their usual brands of tobacco products.
  Interventions: Other: Camel Snus; Other: Cigarettes
- Dual users of moist snuff and cigarettes (Other): Subjects who use both moist snuff and cigarettes as their usual brands of tobacco products.
  Interventions: Other: Moist Snuff; Other: Cigarettes
- Cigarette smokers (Other): Subjects for whom cigarettes is their usual brand of tobacco product.
  Interventions: Other: Cigarettes
- Non-tobacco users (Other): Subjects who do not use tobacco products.
  Interventions: Other: No tobacco usage

INTERVENTIONS:
Other: Moist Snuff — Moist Snuff product
  Arms: Dual users of moist snuff and cigarettes; Moist Snuff users
Other: Camel Snus — Camel Snus product
  Arms: Camel Snus users; Dual users of Camel Snus and cigarette
Other: Cigarettes — Cigarette product
  Arms: Cigarette smokers; Dual users of Camel Snus and cigarette; Dual users of moist snuff and cigarettes
Other: No tobacco usage — No tobacco usage
  Arms: Non-tobacco users

SUMMARY:
This is a multicenter, post market surveillance study designed to evaluate biomarkers of tobacco exposure and effect, health status measurements, and tobacco product usage patterns in subjects who are natural adopters of cigarettes and/or smokeless tobacco. Non tobacco users will serve as a non use comparison group. This study is unblinded by necessity due to the very different visual appearance of the subject's Usual Brand (UB) of tobacco product(s).

DETAILED DESCRIPTION:
A total of approximately 320 subjects will be enrolled in parallel in one of the following 6 cohorts based on tobacco usage:

* Exclusive moist snuff users (n=50)
* Exclusive Camel SNUS users (n=50)
* Dual users of Camel SNUS and cigarettes (n=50)
* Dual users of moist snuff and cigarettes (n=50)
* Exclusive cigarette smokers (n=40 males and 20 females)
* Non tobacco users (n=40 males and 20 females)

The study duration will be 5.5 weeks or less, depending upon the study procedures required for the subject's specific cohort. The study duration includes screening up to 35 days prior to clinic check in (Day 1) and a 2 day confinement period of approximately 24 hours (Day 1 and Day 2). Subjects will be discharged in the morning on Day 2.

At the Initial Screening Visit, clinical study staff will perform screening assessments. Tobacco users will be instructed to provide a sufficient supply of their UB product(s) for use during pre-clinic procedures (i.e., pre-clinic used tobacco product collections) and for use during clinic confinement.

Prior to checking in for clinic confinement, subjects will return to the clinic for a Pre-Enrollment Outpatient Visit to assess enrollment eligibility related to the safe completion of triplicate spirometry and to pick up used tobacco product collection kits and/or urine collection containers for pre-clinic collection procedures. Within 14 days prior to clinic admission, subjects will be instructed, depending on their tobacco cohort, to continue smoking and/or using Camel SNUS or moist snuff at their normal rates and to collect their used cigarette butts (1 day collection) and/or used snus pouches (7 day collection), and retain the labeled snuff containers (1 day usage). Subjects will turn in their used tobacco product collections upon clinic check in.

Subjects will report to the clinical research unit in the morning on Day 1 for baseline testing, confirmation of continued study eligibility, check in of their UB tobacco product(s), and return of their urine collection containers and used tobacco product collections. Subjects will be allowed to use their UB tobacco product(s) ad libitum; tobacco products will be stored by clinic staff and will be dispensed subsequent to subject request, as allowed during scheduled study procedures (i.e., questionnaires, spirometry, carboxyhemoglobin, 6MWT [six-minute walk test]). Each UB product usage will be recorded. At approximately 2200, fasting (from all food and drink except water) and tobacco abstention will begin. Subjects must agree to remain abstinent for approximately 8-10 hours and until all Day 2 fasting procedures (i.e., samples for biomarkers of tobacco effect and exposure) have been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form.
2. Male or female subjects at least 19 years of age.
3. Able to safely perform all study procedures, as determined by the site Investigator.
4. Willing to perform all study procedures and to consume only the meals/snacks provided while confined to the clinic.
5. Agree to not use drugs of abuse over the course of the study, and test negative for drugs of abuse.
6. Test negative for breath alcohol (by breathalyzer).
7. For tobacco users: do NOT intend to quit smoking nor intend to quit using oral smokeless tobacco products (STP) leading up to study participation (defined as planning a quit attempt within a month of the Initial Screening Visit).
8. For tobacco users: willing to abstain from tobacco use for up to 10 hours during overnight confinement in the clinic.
9. Able to read, understand, and complete questionnaires in English.
10. Meet cohort specific requirements as follows:

    * Moist Snuff Users: Must be exclusive moist snuff users of any brand, any style, and any flavor who self-report using on average ≥ 1 can per week for at least 6 months prior to study entry, have an expired carbon monoxide (ECO) level of 0 to 5 ppm, and have a positive urine cotinine screen. Note: Subjects with an ECO level of 6 to 10 ppm may be included upon joint review by the Sponsor and Investigator.
    * Camel SNUS Users: Must be exclusive Camel SNUS users of any variety who self report using on average ≥ 1 tin per week for at least 6 months prior to study entry, have an ECO level of 0 to 5 ppm, and have a positive urine cotinine screen. Note: Subjects with an ECO level of 6 to 10 ppm may be included upon joint review by the Sponsor and Investigator.
    * Dual Camel SNUS/Cigarette Users: Must be dual users of Camel SNUS and allowed commercial filtered tobacco burning cigarettes, using on average ≥ 1 tin of Camel SNUS per week and smoking ≥ 5 cigarettes daily for at least 6 months prior to study entry. The subject's ECO level must be from 5 to 100 ppm, and the urine cotinine screen must be positive.
    * Dual Moist Snuff/Cigarette Users: Must be dual users of moist snuff and allowed commercial filtered tobacco burning cigarettes, using on average ≥ 1 can of snuff per week and smoking ≥ 5 cigarettes daily for at least 6 months prior to study entry. The subject's ECO level must be from 5 to 100 ppm, and the urine cotinine screen must be positive.
    * Cigarette Smokers: Must be exclusive cigarette smokers (of allowed commercial filtered tobacco burning cigarettes) who self-report smoking on average ≥ 10 cigarettes daily for at least 6 months prior to study entry, have an ECO level of 10 to 100 ppm, and have a positive urine cotinine screen.
    * Non Tobacco Users: Must be non tobacco users for at least 12 months prior to study entry with an ECO level of 0 to 5 ppm, and have a negative urine cotinine screen. Note: Subjects with an ECO level of 6 to 10 ppm may be included upon joint review by the Sponsor and Investigator.

Exclusion Criteria:

1. Use of any type of non-tobacco nicotine-containing product/device (e.g., electronic cigarette) or any nicotine replacement therapy (e.g., nicotine patch, nicotine gum, nicotine spray, nicotine inhaler or nicotine lozenge) within 6 months prior to study entry or during the study.
2. Unable to safely perform the study procedures, as determined by the site Investigator. In general, subjects with any of the conditions listed below will be excluded unless individually approved by the Medical Monitor.

   1. Uncontrolled hypertension (blood pressure > 170/110 mmHg at the Initial Screening Visit).
   2. Unstable coronary artery disease (Class III-IV angina).
   3. Decompensated (Class III-IV) congestive heart failure.
   4. Morbid obesity (body mass index [BMI] ≥ 40 kg/m2).
   5. Uncontrolled diabetes (HgbA1c > 9.0).
   6. Pulmonary disease requiring oxygen therapy or preventing 6 minutes of steady ambulation or preventing completion of triplicate spirometry.
   7. Reduced mobility that impairs satisfactory completion of the 6MWT (six minute walk test), such as:

   i. Clinically significant arthritis of the knee or hip.

   ii. Claudication with walking 6 minutes or less.

   iii. Clinically significant ambulation impairment as sequelae of cerebrovascular accident (CVA), sciatica, peripheral nervous disease, or myopathy.

   iv. Imbalance or other gait disorder requiring assistance of a cane or walker to ambulate.
3. Have a resting heart rate (after being seated for at least 5 minutes) of > 120 beats per minute (bpm).
4. Had a myocardial infarction within the month prior to the Initial Screening Visit through enrollment into the study.
5. Have self reported or clinical indications of psychiatric disorders deemed clinically significant by the site Investigator.
6. Unwilling to perform the study procedures.
7. For females: intend to get pregnant during study period, or are currently pregnant or breast feeding.
8. For cigarette- and dual-users:

   1. use of any charcoal-filtered cigarette (i.e., brands such as Lark, Kent, etc., with the word "charcoal" on the package),
   2. use of any crush-capsule cigarette (such as Camel Crush or Pall Mall Crush), or
   3. use of any non tobacco burning cigarette, including tobacco heating cigarettes (such as Eclipse, Accord, etc.) or electronic cigarettes (e-cigarettes such as Smoking Anywhere, Gamucci, NJOY, etc.).
9. For tobacco users: express an interest in quitting smoking or using oral smokeless tobacco (defined as planning a quit attempt within a month of the Initial Screening Visit).
10. Have participated in a clinical study and/or received an investigational product within 30 days of the Initial Screening Visit.
11. Meet cohort specific exclusions as follows:

    * Moist Snuff Users: For 6 months prior to the study through Day 1, the use of any other tobacco- or nicotine-containing product or device other than moist snuff (of any brand, style, and flavor), including tobacco-burning cigarettes, tobacco-heating cigarettes, e cigarettes, cigars, pipes, chewing tobacco, dry snuff, snus, etc.; a negative urine cotinine screen; or an ECO greater than 5 ppm (ECO of 6 to 10 ppm may not exclude based upon joint review by the Sponsor and Investigator).
    * Camel SNUS Users: For 6 months prior to the study through Day 1, the use of any tobacco- or nicotine-containing product or device other than Camel SNUS (of any variety), including tobacco-burning cigarettes, tobacco-heating cigarettes, e cigarettes, cigars, pipes, chewing tobacco, dry snuff, moist snuff, other snus brands, etc.; a negative urine cotinine screen; or an ECO greater than 5 ppm (ECO of 6 to 10 ppm may not exclude based upon joint review by the Sponsor and Investigator).
    * Dual Camel SNUS/Cigarette Users: For 6 months prior to the study through Day 1, the use of any tobacco- or nicotine-containing product or device other than Camel SNUS (of any variety) and tobacco burning cigarettes (allowed commercial filtered cigarettes), including tobacco-heating cigarettes, e cigarettes, cigars, pipes, chewing tobacco, dry snuff, moist snuff, other snus brands, etc.; a negative urine cotinine screen; or an ECO less than 5 or greater than 100 ppm.
    * Dual Moist Snuff/Cigarette Users: For 6 months prior to the study through Day 1, the use of any tobacco- or nicotine-containing product or device other than moist snuff (of any brand, style, and flavor) and tobacco burning cigarettes (allowed commercial filtered cigarettes), including tobacco-heating cigarettes, e cigarettes, cigars, pipes, chewing tobacco, dry snuff, snus, etc.; a negative urine cotinine screen; or an ECO less than 5 or greater than 100 ppm.
    * Cigarette Smokers: For 6 months prior to the study through Day 1, the use of any tobacco- or nicotine-containing product or device other than tobacco burning cigarettes (allowed commercial filtered cigarettes), including tobacco-heating cigarettes, e cigarettes, cigars, pipes, chewing tobacco, dry snuff, moist snuff, snus, etc.; a negative urine cotinine screen; or an ECO less than 10 or greater than 100 ppm.
    * Non Tobacco Users: In their lifetime, the use of more than 20 packs of cigarettes; the use of more than 10 cans, tins, or packs of any smokeless tobacco (chewing tobacco, dry snuff, moist snuff, snus); the use of more than 20 cigars; the use of more than 20 pipes of tobacco; the use of any nicotine replacement therapy, the use of any e cigarette, or use of any combination thereof; a positive urine cotinine screen; or an ECO greater than 5 ppm (ECO of 6 to 10 ppm may not exclude based upon joint review by the Sponsor and Investigator).

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2010-02-13 (Actual); Primary Completion 2010-08-14 (Actual); Study Completion 2010-08-14 (Actual)

PRIMARY OUTCOMES:
Urine creatinine | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Urine nicotine and 9 metabolites | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Tobacco specific nitrosamines in urine | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Acrolein metabolite and acrylamide metabolites in urine | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Crotonaldehyde metabolite in urine | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Benzene metabolite in urine | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
1,3 Butadiene metabolites in urine | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Aromatic amines in urine | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Polycyclic aromatic hydrocarbons metabolites in urine | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Thiocyanate in urine | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Urinary mutagen uptake in strains TA98 and YG1024 | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Isoprostanes and metabolites; prostaglandin PGF2alpha in urine | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Blood nicotine and cotinine | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Thiocyanate in blood | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
Carboxyhemoglobin in blood | After 1 day of product usage
  To establish baseline values for tobacco exposure biomarker levels of natural adopters of each product class and of non-tobacco users.
4-Aminobiphenyl hemoglobin adducts in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Amino Acids in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Glycated hemoglobin in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Total cholesterol in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Triglycerides in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Low density lipoprotein cholesterol in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
High density lipoprotein cholesterol in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Very low density lipoprotein cholesterol in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Apolipoprotein A1 in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Apolipoprotein A2 in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Apolipoprotein B100 in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Lipoprotein(a) in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Oxidized low density lipoprotein in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Folate in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Fibrinogen in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Tissue inhibitor of metalloproteinase 1 in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
hsC-reactive protein in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
alpha-1-antitrypsin in blood | After 1 day of product usage
  To establish baseline values for tobacco effect biomarker levels of natural adopters of each product class and of non-tobacco users.
Tar (mg/day) and nicotine (mg/day) from subject's in-clinic cigarette use OR nicotine (mg/day) from subject's in-clinic snus use | After 1 day of product usage
  To establish baseline values for mouth-level exposure of natural adopters for the product classes of cigarettes and snus.
Functional capacity of subjects completing a 6 Minute Walk Test (6MWT) as assessed by the Dyspnea Modified Borg Scale, pre- and post-6MWT. | After 1 day of product usage
  To establish baseline values for health status of natural adopters of each product class and of non-tobacco users.
Functional capacity of subjects completing a 6 Minute Walk Test (6MWT) as assessed by the Overall Fatigue Modified Borg Scale, pre- and post-6MWT. | After 1 day of product usage
  To establish baseline values for health status of natural adopters of each product class and of non-tobacco users.
Functional capacity of subjects completing a 6 Minute Walk Test (6MWT) as assessed by heart rate (beats/minute), pre- and post-6MWT. | After 1 day of product usage
  To establish baseline values for health status of natural adopters of each product class and of non-tobacco users.
Functional capacity of subjects completing a 6 Minute Walk Test (6MWT) as assessed by oxygen saturation (% SpO2), pre- and post-6MWT. | After 1 day of product usage
  To establish baseline values for health status of natural adopters of each product class and of non-tobacco users.
Functional capacity of subjects completing a 6 Minute Walk Test (6MWT) as assessed by spirometry (FEV1 % predicted), pre- and post-6MWT. | After 1 day of product usage
  To establish baseline values for health status of natural adopters of each product class and of non-tobacco users.
Functional capacity of subjects completing a 6 Minute Walk Test (6MWT) as assessed by spirometry (FEV1 /FVC ratio), pre- and post-6MWT. | After 1 day of product usage
  To establish baseline values for health status of natural adopters of each product class and of non-tobacco users.
Current self-reported health status as measured by the Fagerström Test for Nicotine Dependence. | After 1 day of product usage
  To establish baseline values for health status of natural adopters of each product class and of non-tobacco users.
Current self-reported health status as measured by the Smoking Cessation Quality of Life Questionnaire (SCQoL, inclusive of the Short Form Health Survey [SF-36v2]). | After 1 day of product usage
  To establish baseline values for health status of natural adopters of each product class and of non-tobacco users.
Current self-reported health status as measured by the American Thoracic Society Division of Lung Disease Questionnaire (ATS-DLD-78-A). | After 1 day of product usage
  To establish baseline values for health status of natural adopters of each product class and of non-tobacco users.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbette Jones, DrPH, Study Director — RAIS
Locations (6):
- United States (6):
  - Avail Clinical Research, DeLand, Florida
  - Comprehensive Clinical Development, Inc., Miramar, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Central Kentucky Research Associates (CKRA), Lexington, Kentucky
  - MetaClin Research, Inc., Austin, Texas
  - Community Clinical Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: No